CLINICAL TRIAL: NCT05369364
Title: The Combination of Oral Zanubrutinib and High-dose Dexamethasone vs High-dose Dexamethasone as First-line Treatment in Adult Immune Thrombocytopenia: A Multicenter, Randomized, Open-label Trial
Brief Title: The Combination of Zanubrutinib and High-dose Dexamethasone as First-line Treatment in Adult Immune Thrombocytopenia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Navy General Hospital, Beijing (Other); Beijing Aerospace General Hospital (Other); Qilu Hospital of Shandong University (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDDXM-Zan-ITP
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Immune Thrombocytopenia
Keywords: BTK inhibitor; High-dose Dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — zanubrutinib; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zanubrutinib and HD-DXM (Experimental): Dexamethasone 40 mg per day, 4 consecutive days (the 4-day course of dexamethasone was repeated in the case of lack of response by day 10) and Zanubrutinib 80mg qd po, 6 consecutive weeks
  Interventions: Drug: Zanubrutinib; Drug: Dexamethasone
- HD-DXM (Active Comparator): Dexamethasone 40 mg per day, 4 consecutive days (the 4-day course of dexamethasone was repeated in the case of lack of response by day 10)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib 80mg qd po, 6 consecutive weeks
  Other Names: BTK inihibitor
  Arms: Zanubrutinib and HD-DXM
Drug: Dexamethasone — Dexamethasone, iv, 40 mg/d, for 4 days (The 4-day course of dexamethasone was repeated in the case of lack of response by day 10)
  Other Names: HD-DXM

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of zanubrutinib plus high-dose dexamethasone compared to high-dose dexamethasone monotherapy for the first-line treatment of adults with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of patients with ITP in China. Patients were randomized to Zanubrutinib + high-dose dexamethasone and high-dose dexamethasone monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed newly-diagnosed, treatment-naive ITP;
2. Platelet counts <30×10^9/L ;
3. Platelet counts < 50×10^9/L and significant bleeding symptoms (WHO bleeding scale 2 or above);
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit;
2. Received first-line and second-line ITP-specific treatments (eg, steriods, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) ;
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections;
4. Active infection;
5. Maligancy;
6. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia);
7. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period; a history of clinically significant adverse reactions to previous corticosteroid therapy;
8. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 12 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 12-month follow-up

SECONDARY OUTCOMES:
Initial complete response | 1 month
  Initial complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding.
Initial response | 1 month
  Initial response (R) as platelet count more than 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.
Number of patients with bleeding | 12 months
  Number of patients with bleeding complication ( WHO bleeding score).
Number of patients with adverse events | 12 months
  Number of patients with adverse events
Time to response (TTR) | 12 months
  The time from starting treatment to time of achievement of CR or R
Duration of response (DOR) | 12 months
  Duration of response at 12-month follow up
Loss of response | 12 month
  Platelet counts below 100 x 109/L or bleeding (from CR) or platelet counts below 30 x 109/L, less than 2-fold increase of baseline platelet count or bleeding (from R)
Durable response | 6 months
  Platelet count ≥30 X 10^9/L and at least doubling of the baseline count at 6 mo
Early response | 1 week
  Platelet count ≥30 X 10^9/L and at least doubling baseline at 1 wk
Remission | 12 months
  Platelet count >100 X 10^9/L at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, md, Principal Investigator — Peking University People's Hospital